CLINICAL TRIAL: NCT02720549
Title: The Effect of Remote Ischemic Postconditioning on Postoperative Renal Dysfunction in Patients Undergoing Valvular Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2015-1198
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Valvular Heart Disease Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- post-ischemic conditioning group (Experimental)
  Interventions: Procedure: remote ischemic postconditioning
- valvular surgery with bypass group (Placebo Comparator)
  Interventions: Procedure: valvular surgery with bypass

INTERVENTIONS:
Procedure: remote ischemic postconditioning — Remote ischemic postconditioning post group will take a remote ischemic postconditioning with tourniquet in their lower extremity under thigh. The conditioning is 5 minutes of inflation, and 5 minutes of deflation, repeated 3 cycles.
  Arms: post-ischemic conditioning group
Procedure: valvular surgery with bypass — valvular surgery with bypass
  Arms: valvular surgery with bypass group

SUMMARY:
Ischemic reperfusion injury of cardiopulmonary bypass and postoperative renal dysfunction is a common problem which influence poor outcome in subjects undergoing valvular heart surgery. The incidence of postoperative renal dysfunction was reported as high as 7~8% in heart surgery using bypass, and is thought to be caused by ischemia/reperfusion injury. Remote ischemic postconditioning was also reported to be protective for ischemic/reperfusion injury in previous animal studies and stoke patients. Therefore, the investigators are trying to evaluate the clinical effect of remote ischemic postconditioning on postoperative renal dysfunction in subjects undergoing valvular heart surgery with bypass.

ELIGIBILITY:
Inclusion Criteria:

* patients who are undergoing valvular heart surgery
* Adult
* age 19-80

Exclusion Criteria:

* peripheral vascular disease with circulation deterioration
* Renal replacement therapy
* preconditioning medication
* Myocardiac infarction within 3 weeks
* active infective endocarditis
* high dosage steroid therapy
* mental retardation
* unlettered person

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative renal dysfunction using AKIN(acute kidney injury network) criteria | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song JW, Lee WK, Lee S, Shim JK, Kim HJ, Kwak YL. Remote ischaemic conditioning for prevention of acute kidney injury after valvular heart surgery: a randomised controlled trial. Br J Anaesth. 2018 Nov;121(5):1034-1040. doi: 10.1016/j.bja.2018.07.035. Epub 2018 Sep 18. PMID 30336847